CLINICAL TRIAL: NCT05629793
Title: Differential Diagnosis of Persistent COVID-19 by Artificial Intelligence
Acronym: DICOPERIA
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Fundacin Biomedica Galicia Sur (Other)
Collaborators: University of Vigo (Other); Galician South Health Research Institute (Network)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: DICOPERIA
Record Dates: First submitted 2022-11-18; First posted 2022-11-29 (Actual); Last update posted 2022-11-29 (Actual); Status verified 2022-11

CONDITIONS: COVID-19; Fatigue; Distress Respiratory Syndrome; Cognitive Dysfunction; COVID-19 Recurrent; SARS CoV 2 Infection
Keywords: Machine learning; Stress test; Cardiac variability; Voice recording; Skin conductance
MeSH Terms: conditions — COVID-19; Fatigue; Pulmonary Atelectasis; Cognitive Dysfunction

STUDY DESIGN:
Intervention Model Description: Persistent COVID group vs. Recovered COVID group
Who Masked: Investigator
Masking Description: The investigators performing the tests will be blinded to the diagnostic group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Persistent COVID group (Experimental): Patients with persistent COVID will be recruited by the physicians of the Post COVID-19 Multidisciplinary Clinic of the Complexo Hospitalario Universitario de Ourense.
  Interventions: Other: Experimental tests
- Recovered COVID group (Experimental): The controls will be recruited in a matched manner with the clinical sample in age, sex, epidemic wave and vaccination status, from among previously COVID-positive patients cured without sequelae and attended in Primary Care in the Health Centers of A Cuña, Valle Inclán and Novoa Santos in Ourense.
  Interventions: Other: Experimental tests

INTERVENTIONS:
Other: Experimental tests — Walking for 6 minutes, sitting down and getting up from a chair for 1 minute and finally the cold test (Cold pressor) where the hand is introduced for 1 minute in water at 4ºC. The patient will be monitored by means of a Polar H10 chest strap, as used in sports, continuously and 02 saturation, TA and voice (exhalation while saying /a/ and dry cough) will be collected before and after the tests. Finally, skin conductance will be monitored by performing baseline tracing and then control while performing the cold test.

SUMMARY:
The pandemic caused by SARS-CoV-2 infection has resulted, in addition to the well-known acute symptoms, in the emergence of persistent, diffuse and heterogeneous symptoms referred to as persistent COVID.

Common symptoms include fatigue, shortness of breath, and cognitive dysfunction, among others, and result in an impact on daily functioning. Symptoms may be new onset, appear after initial recovery from an acute episode of COVID-19, or persist after the initial illness. Cardiac variability (HRV) was initially used in COVID-19 to predict mortality in the acute setting. Dysautonomia which partly evaluates HRV is frequent in patients with persistent COVID. Several groups have used voice or other respiratory noise analysis for the diagnosis of acute COVID.

Patients in the persistent COVID cohort will be able to be differentiated from an age, sex and vaccination status matched cohort of recovered COVID patients without sequelae by means of a model created by Machine Learning that will be trained using cardiac variability (HRV), skin conductance and acoustic analysis data. The primary objetive will be to obtain a classification algorithm by Machine Learning to differentiate the group of patients with persistent COVID diagnosis from the paired group of recovered COVID patients without sequelae.

DETAILED DESCRIPTION:
This is a validation study of a Machine Learning algorithm for the diagnosis of persistent COVID using clinical diagnosis as the "gold standard". The sample will be composed of post-COVID patients, one group of which developed persistent COVID and another paired with the previous one with cured COVID without sequelae.

ELIGIBILITY:
Persistent COVID group:

Inclusion Criteria:

* Age ≥18 and ≤70 years of age
* Confirmed infection (PCR) with SARS- CoV-2 until 03/28/2022 and thereafter date.
* Symptoms include: fatigue, respiratory distress or cognitive dysfunction, among others.
* Symptoms persist or appear more than 3 months after onset of infection.
* Symptoms last longer than 2 months and are not better explained by another diagnosis.
* Symptoms appeared after initial recovery or persisted since disease debut.
* Symptoms may fluctuate or remit over time.
* Patients have capacity to consent and agree to participate in the study.

Exclusion Criteria:

* Active COVID-19 infection.
* Cardiac arrhythmia, pacemaker carrier.
* Other pathologies with dysautonomia.
* Raynaud's phenomenon.
* Other diseases that may affect exercise capacity or be aggravated by exercise shall also be excluded, such as: Uncontrolled heart failure, severe or symptomatic aortic stenosis, pulmonary edema, acute respiratory failure, recent pulmonary thromboembolism, lower limb thrombosis, infections, thyrotoxicosis, or orthopedic inability to walk.

Recovery COVID group

Inclusion Criteria:

* Age ≥18 and ≤70 years of age
* Confirmed infection (PCR) with SARS- CoV-2 until 03/28/2022 and thereafter date.
* Full functional recovery.
* Follow-up by Primary Care.
* They have not presented three months after the onset of the disease: fatigue, respiratory distress or cognitive dysfunction, among others.
* Patients have capacity to consent and agree to participate in the study.

Exclusion Criteria:

* Active COVID-19 infection.
* Cardiac arrhythmia, pacemaker carrier.
* Other pathologies with dysautonomia.
* Raynaud's phenomenon.
* Other diseases that may affect exercise capacity or be aggravated by exercise such as: uncontrolled heart failure, severe or symptomatic aortic stenosis, pulmonary edema, acute respiratory failure, recent pulmonary thromboembolism, lower limb thrombosis, infections, thyrotoxicosis, or orthopedic inability to walk shall also be excluded.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 136 (Estimated)
Dates: Start 2022-12-14 (Estimated); Primary Completion 2023-11 (Estimated); Study Completion 2023-11 (Estimated)

PRIMARY OUTCOMES:
Differences of the group of patients with a persistent diagnosis of COVID from the age-matched group, sex and vaccination status of patients recovered from COVID without sequelae. | 8 weeks
  Through an algorithm model created by Machine Learning that will be trained using cardic variability (HRV), skin conductance and acoustic analysis data.

SECONDARY OUTCOMES:
Cardiac variability | 8 weeks
  Number of times a contraction of the heart occurs in one minute, expressed in beats per minute, by means of a Polar chest strap, model H10. A baseline recording of 5 minutes duration will be taken, with the patient in a seated position. At the end of each test, recording is continued for 2 minutes to demonstrate the speed and degree of recovery after stress.
Voice recording | 8 weeks
  Sounds produced by the patient at rest and after having performed the stress tests. The patient will be asked to take a deep breath and then pronounce the vowel /a/ in a sustained manner, in a comfortable tone and volume (3 times).
Skin conductance | 8 weeks
  micro Siemens [µS]. By means of the Bitalino electrodermal activity recording system. It will be recorded at rest, during the Cold Pressor test and once it is finished, for at least two minutes, to assess the normalization of the conductivity curve.
6MWT | 8 weeks
  metres/min. The patient will walk the maximum distance they can in 6 minutes.
1minSTST | 8 weeks
  Number of repetitions performed after sitting down and getting up from a chair without supporting the hands as many times as possible for 1 minute..
Cold Pressor test | 8 weeks
  One hand is inserted into a container with water at 4-5ºC for 1 minute. Before and after the test, HRV, BP, and thermal conductance are recorded for 5 and 2 minutes -respectively- while lying supine.

OTHER OUTCOMES:
Age | 8 weeks
  Years
Sex | 8 weeks
  Male, Female
Current treatment | 8 weeks
  Treatment taken by the patient at the time of the study.
Date of PCR + SARS-CoV-2 | 8 weeks
  DD-MMM-YYYY
Epidemic wave | 8 weeks
  Of the 7 waves of COVID-19 that have occurred in Spain, a description will be given of the wave to which the infection of each patient included belonged. First, second, third, fourth, fifth, sixth, seventh, eighth, ninth or tenth wave.
Vaccination status at the time of infection | 8 weeks
  Number of vaccines doses at the time of infection
FVC | 8 weeks
  Is the maximum volume of air exhaled, with the maximum possible effort, starting from a maximum inspiration in ml.
FEV1 | 8 weeks
  The volume of air expelled during the first second of forced expiration in ml.
FEV1/ FVC | 8 weeks
  Expressed as a percentage (%), it indicates the proportion of the FVC that is expelled during the first second of the forced expiratory maneuver.
CO diffusion test | 8 weeks
  To evaluate the transfer of oxygen from the alveolar space to the hemoglobin of the erythrocytes contained in the pulmonary capillaries. Effective alveolar-capillary area available for gas transfer in the lung. (%)

CONTACTS AND LOCATIONS:
Locations (7):
- Spain (7):
  - Complexo Hospitalario Universitario de Ourense, Ourense
  - Health Center Novoa Santos, Ourense
  - Health Center Valle Inclán, Ourense
  - S.S. Computer Engineering (University of Vigo), Ourense
  - Health Center A Cuña, Ourense
  - Galicia Sur Health Research Institute (IISGS) - Hospital Álvaro Cunqueiro, Vigo
  - School of Telecommunication Engineering (University of Vigo), Vigo